CLINICAL TRIAL: NCT00728234
Title: Analysis of Amplitude-Integrated Electroencephalography and Its Predictive Value for Neurodevelopmental Outcome in Preterm Infants Born Below 30 Weeks Gestational Age
Brief Title: Analysis of Correlation of Amplitude-Integrated EEG and Neurodevelopmental Outcome in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Dr.Katrin Klebermass, Univ.Prof.Dr.Manfred Weninger, Medical University Vienna, Department of Pediatrics
Other Study IDs: Klebermass_01
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2008-07

CONDITIONS: Brain Activity; Neurodevelopmental Outcome
Keywords: aEEG; preterm infants; predictive value; outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: all infants born below 30 weeks gestational age at the medical university vienna within the study period (01/2000 - 12/2002)
  Interventions: Device: aEEG recording

INTERVENTIONS:
Device: aEEG recording — weekly recordings with aEEG
  Other Names: 1 - all infants < 30 weeks gestational age

SUMMARY:
The study included analysis of longitudinal recordings of amplitude-integrated EEG (aEEG) tracings on a weekly basis in preterm infants and evaluation of their neurodevelopmental outcome at the age of three years.

Aim of the study was to observe if there is a correlation of the aEEG tracings of the first weeks of life to later neurodevelopmental outcome and to evaluate if aEEG can be used as prognostic tool.

DETAILED DESCRIPTION:
From the first week of life on aEEG-recordings were obtained on a weekly basis and the results of the first eight weeks of life were analyzed for this study.

aEEG-tracings were analyzed with regard to background activity (percentages of continuous and discontinuous patterns), the presence/absence of sleep-wake-cycles and the occurrence of seizure activity. These items where summed up in a score including three grades (normal, moderately and severely abnormal).

The aEEG was recorded as a single channel EEG from biparietal surface disk electrodes using a CFM (CFM 5330, Lectromed Devices Ltd., UK) or the CFM 6000 (Olympic Medical, USA). Assessment of neurodevelopmental outcome was done at three years of age by assessment of the Bayley Scales of Infant Development II (BSID-II) During the study period from January 1st 2000, and December 31st 2002 a total of 284 preterm infants less than 30 weeks´ gestational age were admitted to the neonatal intensive care unit of the Medical University of Vienna. Neurodevelopmental outcome could be obtained in 148/284 infants at the age of three years and these infants therefore fulfilled the inclusion criteria for this study

ELIGIBILITY:
Inclusion Criteria:

* gestational age < 30 weeks

Exclusion Criteria:

* brain malformation
* inborn error of metabolism

Ages: 23 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: inclusion of all preterm infants born below 30 weeks gestational age within the study period at medical university vienna
Sampling Method: Non-Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2000-01; Primary Completion 2002-12 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
amplitude-integrated electroencephalography tracings of the first weeks of life; obtained on a weekly basis | 8-12 weeks

SECONDARY OUTCOMES:
neurodevelopmental outcome at the age of three years assessed by Bayley Scales of Infant Development | three years

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Pollak, MD, PhD, Study Chair — Medical University Vienna, Head of Department of Pediatrics
Locations (1):
- Medical University, Vienna, Austria

REFERENCES:
- [Derived] Klebermass K, Olischar M, Waldhoer T, Fuiko R, Pollak A, Weninger M. Amplitude-integrated EEG pattern predicts further outcome in preterm infants. Pediatr Res. 2011 Jul;70(1):102-8. doi: 10.1203/PDR.0b013e31821ba200. PMID 21436758